CLINICAL TRIAL: NCT05028049
Title: Comparison of Remifentanil-induced Postoperative Hyperalgesia After Gynecological Laparoscopic Surgery Between Patients From the Plain Area and the Plateau Area
Brief Title: Comparison of Remifentanil-induced Postoperative Hyperalgesia Between Patients From Plain Area and Plateau Area
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Guolin Wang, Professor, Tianjin Medical University General Hospital
Other Study IDs: GWang014
Record Dates: First submitted 2021-08-21; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Pain, Postoperative; Anesthesia
Keywords: Remifentanil; Opioid-induced hyperalgesia; Postoperative pain; pain intensity
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Sufentanil; Remifentanil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Sufentanil-analgesia in plain area patients: Sufentanil 0.3 μg/kg is intravenously administrated to maintain intraoperative analgesia in plain area patients.
  Interventions: Drug: Sufentanil injection; Other: plain areas
- Remifentanil-analgesia in plain area patients: Remifentanil 0.3ug/kg/min is intravenously administrated to maintain intraoperative analgesia in plain area patients.
  Interventions: Drug: Remifentanil Hydrochloride; Other: plain areas
- Sufentanil-analgesia in plateau area patients: Sufentanil 0.3 μg/kg is intravenously administrated to maintain intraoperative analgesia in plateau area patients.
  Interventions: Drug: Sufentanil injection; Other: plateau areas
- Remifentanil-analgesia in plateau area patients: Remifentanil 0.3ug/kg/min is intravenously administrated to maintain intraoperative analgesia in plateau area patients.
  Interventions: Drug: Remifentanil Hydrochloride; Other: plateau areas

INTERVENTIONS:
Drug: Sufentanil injection — Sufentanil 0.3 μg/kg is intravenously administrated to maintain intraoperative analgesia
  Other Names: Sufentanil
  Groups: Sufentanil-analgesia in plain area patients; Sufentanil-analgesia in plateau area patients
Drug: Remifentanil Hydrochloride — Remifentanil 0.3ug/kg/min is intravenously administrated to maintain intraoperative analgesia
  Other Names: Remifentanil
  Groups: Remifentanil-analgesia in plain area patients; Remifentanil-analgesia in plateau area patients
Other: plain areas — Patients should be long staying residents in plain areas (altitude level below 1,000 meters above sea level)
  Groups: Remifentanil-analgesia in plain area patients; Sufentanil-analgesia in plain area patients
Other: plateau areas — Patients should be long staying residents in plateau areas (altitude level>3000 meters above sea level)
  Groups: Remifentanil-analgesia in plateau area patients; Sufentanil-analgesia in plateau area patients

SUMMARY:
Purpose:

1. To compare the incidence of postoperative hyperalgesia induced by remifentanil in patients undergoing gynecological laparoscopic surgery in plateau and plain areas
2. To compare the peri-operative analgesic requirements of patients in plain and plateau areas

DETAILED DESCRIPTION:
Our research group has been committed to the research of remifentanil-induced hyperalgesia for a long time. In the previous study, it was found that intraoperative infusion of remifentanil (0.3ug/kg•min) >1h can lead to remifentanil-induced hyperalgesia and the incidence rate is relative high in the plain area. Due to the long-term low pressure and hypoxia of people living in plateau areas, a series of changes will occur in the respiratory and circulatory systems, and their anesthesia management needs to be adjusted accordingly. However, there is no relevant research on whether or not hyperalgesia occurs in people in plateau areas (altitude level >3000 meters). Therefore, this study hopes to compare the incidence and degree of remifentanil-induced hyperalgesia after gynecological laparoscopic surgery in plain areas and plateau areas.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is scheduled to undergo gynecological laparoscopic surgery under a short general anesthesia of less than 2 hours
2. Subject's American Society of Anesthesiologists physical status is I-II.
3. The subject's parent/legally authorized guardian has given written informed consent to participate.
4. Patients in plateau areas are long staying residents in above 3000 meters above sea level for enrollment, while patients in plain areas are long staying residents below 1000 meters above sea level.

Exclusion Criteria:

1. Subject has a diagnosis of renal or liver failure.
2. Subject has a diagnosis of Insulin dependent diabetes.
3. Subject is allergy and contraindication to any drugs used during general anesthesia.
4. Subject has a history of chronic pain, a history of alcohol or opioid abuse, pre-existing therapy with opioids, intake of any analgesic drug within 48 hours before surgery.
5. Subject has any contraindication for the use of patient-controlled analgesia (PCA).
6. Subject is pregnant or breast-feeding.
7. Subject is obese (body mass index >30kg/m2).

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — We selected female patients which will receive gynecological laparoscopic surgery
Study Population: Patients in plateau areas are long staying residents in above 3000 meters above sea level for enrollment, while patients in plain areas are long staying residents below 1000 meters above sea level.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-08-30 (Estimated); Primary Completion 2021-12-15 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Mechanical Hyperalgesia Threshold on the Dominant Inner Forearm | 48 hours after surgery
  The mechanical hyperalgesia threshold was defined as the lowest force (g) necessary to bend a Von Frey filament, which was perceived to be painful by the patient and measured by Von Frey filament after surgery

SECONDARY OUTCOMES:
Pain Score (NRS) | 48 hours after surgery
  The pain score at rest or after movement was evaluated by pain 11-point numerical rating scale (NRS): 0 = no pain, 10= greatest imaginable pain.
Normalized Area of Hyperalgesia Around the Incision | 48 hours after surgery
  The skin around the incision is stimulated in steps of 5 mm at intervals of 1 s starting outside of the hyperalgesic area in the direction of the incision. The distance from the incision to the first point where a'painful', 'sore' or 'sharper' feeling occurred is measured and noted. This measurement is repeated at predefined radial lines around the incision. To eliminate the variable length of incision, this length is subtracted from the longer diameter leaving four radial distances from the end and from the middle of the incision. The normalized area of hyperalgesia is calculated by summing up the areas of the remaining four triangles measured by and Von Frey filament.
Mechanical hyperalgesia threshold around the incision | 48 hours after surgery
  The mechanical hyperalgesia threshold was defined as the lowest force (g) necessary to bend a Von Frey filament, which was perceived to be painful by the patient and measured by Von Frey filament.
Time of First Postoperative Analgesic Requirement | 1 hour after surgery
  First postoperative pain (NRS≥5) is initially controlled by titration of Hydromorphone.
Total Dose of First Postoperative Analgesic Requirement | 1 hour after surgery
  First postoperative pain (NRS≥5) is initially controlled by titration of Hydromorphone.
Cumulative Hydromorphone Consumption | 48 hours after surgery
  Each patient was administered analgesics using a PCA (Patient-controlled analgesia) pump containing Hydromorphone (200μg) in normal saline at a total volume of 100 ml after leaving PACU (Postanesthesia care unit). This device was set to deliver a basal infusion of 2 ml/h and bolus doses of 0.5 ml with a 15-min lockout period. Hydromorphone cumulative consumption is recorded 48 hours postoperatively
Occurrence of Side Effects | 48 hours after surgery
  Occurrence of side effects: nausea, vomiting, dizziness, headache, shivering, pruritus

CONTACTS AND LOCATIONS:
Overall Officials: Guolin Wang, MD, Study Director — Tianjin Medical University General Hospital
Locations (2):
- China (2):
  - Gannan Tibetan Autonomous Prefecture People's Hospital, Hezuo, Gansu
  - Tianjin Medical University General Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No